CLINICAL TRIAL: NCT06280586
Title: Effectiveness of a Multimodal and Multidisciplinary Intervention (ESPAI-Fragility) in the Prevention of Sarcopenia, Frailty and Functional Decline in Pre-frail Elderly in the Community. Randomized Controlled Clinical Trial.
Brief Title: Effectiveness of Intervention in Prevention of Sarcopenia, Frailty and Functional Decline in Pre-frail Community Elderly
Acronym: ESPAI-F
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Principal Investigator, Mateu Serra Prat, MD PhD, Consorci Sanitari del Maresme
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 44/21
Record Dates: First submitted 2023-12-22; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Muscle Strengh; Frailty; Sarcopenia
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual clinical practice
- Intervention (Experimental): * bimonthly personalized follow-up with the appropriate specialists (5 in a year) i
  * a program of group activities (6 sessions in a year) with a monitor with the aim of reinforcing adherence to the study intervention and adapting it to the circumstances and the physical, personal and social reality around each participant. The sessions will last approximately one hour and will cover:
    * General dietary and hydration recommendations and dietary recommendations for people at risk of malnutrition
    * Dietary and physical exercise recommendations in obese elderly
    * General physical exercise recommendations in the elderly and physical exercise recommendations in the elderly with sarcopenia
    * Physical exercise recommendations for the elderly at risk of falls.
    * Medication management and social resources for the elderly in Mataró.
  Interventions: Other: Multidisciplinary intervention

INTERVENTIONS:
Other: Multidisciplinary intervention — * bimonthly personalized follow-up with the appropriate specialists (5 in a year) i
  * a program of group activities (6 sessions in a year) with a monitor with the aim of reinforcing adherence to the study intervention and adapting it to the circumstances and the physical, personal and social reality around each participant. The sessions will last approximately one hour and will cover:
    * General dietary and hydration recommendations and dietary recommendations for people at risk of malnutrition
    * Dietary and physical exercise recommendations in obese elderly
    * General physical exercise recommendations in the elderly and physical exercise recommendations in the elderly with sarcopenia
    * Physical exercise recommendations for the elderly at risk of falls.
    * Medication management and social resources for the elderly in Mataró.
  Arms: Intervention

SUMMARY:
Frailty is a geriatric syndrome characterized by a decrease in the function of various organs and systems that leads to a greater risk of suffering from diseases or disabilities. Frailty is usually accompanied by weight loss, loss of strength, slowing of walking speed, fatigue and poor physical activity. Frail people have more difficulty in carrying out the usual activities of daily life and a greater risk of needing help to be able to do them.

The aim of this study is to evaluate the safety and effectiveness of an intervention based on the control of chronic diseases, a good use of medicines, diet, physical exercise and good social support, in the prevention . of frailty in old people who are at risk of frailty.

These criteria for participating in the study are why we invite you to participate. Your participation is voluntary. Your decision to participate or not in the study will not affect the medical care you may need. Before making a decision, read this information sheet carefully and ask the person who informs you the questions you want.

In the study there will be two groups, one will receive the study intervention and the other will not receive any special treatment (we call it the control group). The assignment of each individual to one group or the other will take place once you have decided to participate. This assignment will be made at random so that neither you nor your doctor can know "a priori" which group you will be in.

DETAILED DESCRIPTION:
General objective:

To assess the effectiveness and safety of a multimodal and multidisciplinary intervention in the prevention of sarcopenia, frailty and functional decline in pre-frail community elders aged 70 years or older.

Specific objectives:

1. Evaluate the effect of the study intervention in the medium term (1 year) in terms of prevention or improvement of:

   1. Muscle strength, muscle mass and sarcopenia,
   2. The fragility
   3. Functional capacity (and/or dependence), balance and the risk of falls
   4. Nutritional status
   5. The quality of life
   6. The consumption of health resources in pre-frail community elders 70 years or older.
2. To evaluate the safety of the mid-term study intervention (1 year) in pre-frail community elders aged 70 years or older.

Secondary objectives:

1. Assess the degree of adherence to the study intervention.
2. Evaluate the factors related to good adherence to the study intervention.
3. Describe the main characteristics of pre-frail community elders and analyze the factors associated with sarcopenia and functional impairment in the study population (cross-sectional analysis).
4. Describe the survival of the study sample and find out what the main determinants are (longitudinal analysis).

ELIGIBILITY:
Inclusion Criteria:

* Men or women 70 years of age or older at the time of recruitment
* That they meet pre-frail phenotype criteria according to L. Fried's criteria
* That they give their written informed consent to participate in the study.

Exclusion Criteria:

* Severe dementia (GDS>3)
* Other neurodegenerative diseases (Parkinson's disease)
* Neuromuscular diseases
* Serious psychiatric illness that, at the doctor's discretion, prevents good compliance with the study intervention
* Active cancer
* Life expectancy of less than 6 months
* Institutionalized patient
* Unstable ischemic heart disease, uncontrolled arrhythmias, dissecting aortic aneurysm, severe aortic stenosis, uncontrolled arterial hypertension (>180/100mmHg), or severe heart failure.
* Acute diseases or acute or poorly controlled chronic diseases
* Bone fractures in the last 3 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Mass | baseline, 6 months and 12 months
  Bioimpedance
Muscle strength and/or Muscle function | baseline, 6 months and 12 months
  Isokinetic
Sarcopenia | baseline, 6 months and 12 months
  EWGSOP2 description
Frailty | baseline, 6 months and 12 months
  L Fried Criteria

SECONDARY OUTCOMES:
Functional Capacity 1 | baseline, 6 months and 12 months
  Barthel index
Functional Capacity 2 | baseline, 6 months and 12 months
  Lawton index
Functional Capacity 3 | baseline, 6 months and 12 months
  Timed up and go test
Functional Capacity 4 | baseline, 6 months and 12 months
  SPPB
Functional Capacity 5 | baseline, 6 months and 12 months
  Unipodal test
Functional Capacity 6 | baseline, 6 months and 12 months
  Walking speed mesured by looking time to walk 4.6 meters

CONTACTS AND LOCATIONS:
Overall Officials: Mateu Serra-Prat, MD PhD, Principal Investigator — Fundació Privada Salut del Consorci Sanitari del Maresme
Locations (2):
- Spain (2):
  - Consorci Sanitari del Maresme, Mataró, Barcelona
  - Mateu Serra-Prat, Mataró, Barcelona

IPD SHARING:
Plan to Share IPD: No